CLINICAL TRIAL: NCT03169270
Title: Muscular Adaptations After Endurance Exercise Training in Patients With COPD
Brief Title: Muscular Training-induced Changes in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Josep Roca, Consultor senior, Hospital Clinic of Barcelona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Muscle-COPD
Record Dates: First submitted 2017-05-23; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Chronic Obstructive Pulmonary Disease; Healthy
Keywords: Exercise training; Muscle dysfunction; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPD training group (Experimental): COPD were required to be clinically stable at the time of study without episodes of exacerbation or oral steroid treatment in the previous four months. All COPD patients were on bronchodilators and inhaled corticosteroids. No patient presented severe co-morbidities. The intervention consists in an 8-week programe of exercise training.
  Interventions: Other: Exercise training
- Healthy training group (Active Comparator): Healthy sedentary age-matched subjects were recruited from the outpatients' clinics of our hospital. The intervention consists in an 8-week programe of exercise training.
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — All subjects performed a supervised 8-week, 5 days-week of endurance exercise training program in cycle-ergometer Each session included 5 minutes of warm-up and cool-down pedalling at 30% of peak work-rate (WR) and 50 minutes of interval training. The interval training combined 2 minutes of high-intensity pedalling and 3 minutes of active rest. Work-rate progress during the 8-week period was tailored on individual basis, according to subjects' symptoms, to maximize the training effect. During the first 2 weeks, high intensity pedalling interval was at least 70% of peak WR and active rest interval was at least 40% of peak WR. Thereafter, work-rate was increased by approximately 5% every week up to a maximum of 100% of peak WR during the last 2 weeks for the high intensity period and 50% of peak WR for the active rest. The cycling rate during the sessions was maintained at 60-70 rpm.

SUMMARY:
The current protocol is developed in the context of a large Research and Innovation (R&I) program aiming the promotion of daily life physical activity in chronic patients registered at clinicaltrials.gov (NCT02976064) and approved by the ethical committee of the Hospital Clinic de Barcelona (HCB/2016/0883). The project is partly supported by the Smart Innovation Strategies promoted by the EU Commission (COMRDI15-1-0016). Specifically, the protocol uses retrospective information collected between 2005-2008 as part of the EU project Biobridge (LSHG-CT-2006-037939).

The aims of the current analysis of the retrospective information are 1) to assess training-induced changes in muscle oxygen saturation (StO2) assessed by near-infrared spectroscopy (NIRS) during constant-work rate cycling exercise (CWRE) as a useful marker of the effects of training at limb muscle level in patients with chronic obstructive pulmonary disease (COPD), and 2) to further explore underlying mechanisms of skeletal muscle dysfunction as a characteristic systemic effect of COPD, potentially modifiable with preventive interventions as endurance muscle training.

Methods: Incremental exercise (VO2 peak) and CWRE at 70% baseline peak work rate, before and after 8-week of endurance exercise training, were done in healthy sedentary subjects and COPD patients. NIRS was used to assess StO2 in the left "vastus internus" during the CWRE (before an after training program) (objective 1); and blood samples and muscle biopsies of the quadriceps were obtained at rest (before an after training program) (objective 2).

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis following GOLD criteria (FEV1/FVC post-broncodilator <0,7)
* Clinical stability for at least 3 months

Exclusion Criteria:

* Age <45 years
* Any active cancer
* Comorbidities which carry high-level of handicap
* Other respiratory disease than COPD
* No sign of informed consent

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-11 (Actual); Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Muscle oxygen saturation (StO2) | Baseline - 8 weeks
  Near-infrared spectroscopy (NIRS)
Skeletal muscle dysfunction | Baseline - 8 weeks
  Quadriceps muscle biopsies

SECONDARY OUTCOMES:
Maximal cardiopulmonary response to exercise training | Baseline - 8 weeks
  Incremental exercise test
Submaximal cardiopulmonary response to exercise training | Baseline - 8 weeks
  Constant work rate exercise test (CWRE)
Systemic effects of COPD | Baseline - 8 weeks
  Blood sample

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tenyi A, Cano I, Marabita F, Kiani N, Kalko SG, Barreiro E, de Atauri P, Cascante M, Gomez-Cabrero D, Roca J. Network modules uncover mechanisms of skeletal muscle dysfunction in COPD patients. J Transl Med. 2018 Feb 20;16(1):34. doi: 10.1186/s12967-018-1405-y. PMID 29463285